CLINICAL TRIAL: NCT01999621
Title: Determinants of Intensity of Care of Lung Cancer Patients With Organ Failure
Acronym: CBP-DO
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-16
Record Dates: First submitted 2013-10-15; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Lung Cancer
Keywords: organ failure; intensive care; palliative care; patient's wishes
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung cancer: Each lung cancer patient with organ failure, admitted in emergency, thoracic oncology or directly in ICU

SUMMARY:
Investigators will evaluate determinants of the patients' care type : palliative, medical or intensive care. The place of patient or family on care's decision will be noticed. Investigators will evaluate 3 month-survival and patients' feelings (visit with a psychologist) according to type of care they benefited.

DETAILED DESCRIPTION:
Two hundred patients have to be enrolled in 2 years in the Grenoble Teaching Hospital and in the Saint Louis hospital in Paris between November 2010 and November 2012. Each lung cancer patient with at least one organ failure, admitted in emergency, thoracic oncology or directly in ICU will be included.

The objectives are to identify patients' characteristics associated with proposition for intensive care unit admission and those associated with the decision of intensive care unit admission.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* Organ failure

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each lung cancer patient with organ failure, admitted in emergency, thoracic oncology or directly in ICU will be included
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Identify an association between patients' characteristics and proposition for intensive care unit admission. | at day 0
  univariate and multivariate logistic regression

SECONDARY OUTCOMES:
Identify an association between patients' characteristics and decision of intensive care unit admission among patients proposed for ICU admission | at day 0
  univariate and multivariate logistic regression

OTHER OUTCOMES:
identify patients' characteristics associated with survival | up to 4 months after the last inclusion
  Cox' model
patients' feelings according to intensity of care they received | at 3 months
  hospital anxiety and depression scale, SF-36 scale and Impact of Event Scale-R and a visit with a psychologist

CONTACTS AND LOCATIONS:
Overall Officials: TIMSIT Jean-François, PU/PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France